CLINICAL TRIAL: NCT03634319
Title: Early Evaluation of the Brown Glaucoma Implant in Patients Refractory to Drug Therapy in the European Union
Brief Title: Early Evaluation of the Beacon Aqueous Microshunt in Patients Refractory to Drug Therapy in the European Union
Acronym: EARLY BIRD EU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Significant risks (e.g., infection, endothelial cell loss) and high rate of channel plugging associated with product use.
Sponsor: MicroOptx (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4004-22
Record Dates: First submitted 2018-06-25; First posted 2018-08-16 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: The Beacon Aqueous Microshunt is an implantable device designed to lower intraocular pressure (IOP) in glaucoma patients by shunting aqueous humor from the anterior chamber of the eye to the surface of the eye.
  Because there are no physiologic sources of outflow resistance, the device can be engineered to target an IOP that is low enough to halt the progression to blindness in a patient suffering from glaucoma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Beacon Aqueous Microshunt — The Beacon Aqueous Microshunt is an implantable device designed to lower intraocular pressure (IOP) in glaucoma patients by shunting aqueous humor from the anterior chamber of the eye to the surface of the eye.
  Because there are no physiologic sources of outflow resistance, the device can be engineered to target an IOP that is low enough to halt the progression to blindness in a patient suffering from glaucoma.

SUMMARY:
This is prospective, non-randomized, single-arm study to assess the safety and effectiveness of lowering intraocular pressure with the Beacon Aqueous Microshunt. A total of 65 subjects will be enrolled at five centers. The primary endpoint will be assessed at 12 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 22 years and older.
2. Diagnosed with mild, moderate or severe open-angle glaucoma (OAG).
3. Best corrected vision acuity 20/25 or worse in the study eye.
4. Inadequate medical control of IOP, or target IOP not reached with intraocular pressure in the study eye greater than or equal to 20 mmHg.
5. At least two contiguous clock hours of intact conjunctiva near the limbus between clock hours of 09:00 and 03:00 in the study eye.
6. Adequate space in the anterior chamber of the study eye sufficient to support implant with the BAM, defined as two contiguous clock hours of scleral spur visualization via gonioscopy, without compression, in the superior 180 degrees of the anterior angle.
7. Any IOP-lowering medications should be stabilized at least 30 days prior to baseline measurements.
8. Able and willing to comply with protocol requirements.
9. Able to understand and sign the Informed Consent form.

Exclusion Criteria:

1. Active Neovascular Glaucoma in the study eye.
2. Pigmentary Glaucoma in the study eye.
3. Pseudoexfoliative Glaucoma in the study eye.
4. Any eye disease associated with the formation of free-floating material or tissue in the anterior chamber of the eye.
5. Corneal conditions in the study eye that may inhibit normal incisional healing (e.g. Fuch's dystrophy) or impair visualization of the implant inside the anterior chamber.
6. Anticipated need for ocular surgery within one year in the study eye.
7. Contact lens use in the study eye.
8. Clinically significant inflammation or infection in the study eye within 60 days prior to the preoperative visit (e.g., blepharitis, conjunctivitis, keratitis, uveitis, herpes simplex infection) or any systemic infection. For purposes of this study, clinically significant is considered any such condition requiring prescription therapy.
9. Other clinical conditions:

   1. Poorly controlled diabetes (Type I or Type II) as determined by HbA1c >8.
   2. Cancer requiring treatment during the duration of the study.
   3. Any drugs (e.g.: immunosuppressive drugs) or co- morbidity that might inhibit wound healing.
10. Participation in any other clinical trial during participation in this trial.
11. Life expectancy <1 year.
12. Clinically significant macular degeneration in the study eye.
13. Patients who have undergone surgery in the trial eye within the last 6 months.
14. Planned combined cataract surgery.

If both eyes of a prospective trial participant are eligible, the eye with the highest intraocular pressure will be selected for implant.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2023-01-08 (Actual)

PRIMARY OUTCOMES:
Reduction in IOP | 12 Months
  Overall responder rate, with responder defined as a subject with a diurnal intra-ocular pressure equal to or lower than the individually pre-determined target IOP.
Adverse Event Rate | 12 Months
  Rate of all AEs

SECONDARY OUTCOMES:
Mean Change from Baseline in IOP | 12 Months
  Change in IOP at follow-up compared to baseline
Responder Rate for 20% reduction | 12 Months
  Defined as a subject achieving at least 20% reduction from baseline in IOP
Reduction in IOP lowering medication | 12 Months
  Change in number of medications at follow-up compared to baseline

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Eye Hospital, Bochum
  - Universitatsklinikum Schleswig-Holstein, Lübeck

IPD SHARING:
Plan to Share IPD: No